CLINICAL TRIAL: NCT03078673
Title: Motor Skill- and Strength Training; Importance for Technique, Work Economy and Time Performance in Cross Country Poling
Brief Title: Cross Country Poling Specific Motor Skill- and Strength Training.
Acronym: CPMST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South-Eastern Norway (Other)
Collaborators: The Norwegian Olympic Sports Center (Olympiatoppen) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CPMST
Record Dates: First submitted 2016-05-30; First posted 2017-03-13 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: Cross country poling, motor skill, strength training
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor skill training (Experimental): training intervention. Poling specific indoor motor skill exercises performed 3 times pr week for 10 weeks in addition to regular training
  Interventions: Other: training intervention, motor skill training
- Maximal strength training (Experimental): training intervention. Maximal strength exercises performed 3 times pr week for 10 weeks in addition to regular training
  Interventions: Other: training intervention, maximal strength training
- Control group (Experimental): Only regular training
  Interventions: Other: control group

INTERVENTIONS:
Other: training intervention, motor skill training — cross country specific motor skill strength training
  Arms: Motor skill training
Other: training intervention, maximal strength training — general maximal strength training
  Arms: Maximal strength training
Other: control group — regular training
  Arms: Control group

SUMMARY:
Will motor skill- and/or strength training affect technique, work economy and time performance in cross-country poling? Competitive cross-country skiers (age 16- 30) will perform a 10 weeks training intervention. They will be randomized in one of the following three groups: poling specific motor skill training 3 times per week in addition to their regular training, maximal strength training 3 times per week in addition to their regular training and a control group who only perform their regular training. Pre- and post intervention, all participants will perform tests in VO2max (running), VO2max (poling), work economy (poling), video and inertial measurement unit (IMU) analyzes of poling technique, time performance test (poling), motor skill tests and maximal strength tests.

DETAILED DESCRIPTION:
Motor Skill- and Maximal Strength Training; Importance for Technique, Work Economy and Time Performance in Cross Country Poling Purpose The relative use of poling in classic cross-country skiing has increased over the last years. (Danielsen et al 2015). As a result of this poling performance has become increasingly important for over all classic cross-country skiing performance. Poling performance with best possible technical skills, implying high velocity with a least possible energy cost (C) should thus be beneficial. Previous research (Østerås et al 2002) has shown improved work economy in poling after maximal strength training (MST). To the investigators knowledge, the effect of motor skill training (MOT) on C has not previously been investigated. In this study MOT and MST will therefore be investigated (in two different groups of cross-country skiers), how they may affect poling technique, C, lactate threshold (LT) and poling performance. The results from this study may give further insight and knowledge in scientific based training practice.

The purpose of this study is thus to investigate if:

1. MOT results in technical changes in poling?
2. MST results in technical changes in poling?
3. MOT improves C in poling?
4. MST improves C in poling?
5. changes in 1-4 improves time performance in poling?

In order to investigate this, competitive cross-country skiers (age 16- 30) will perform a 10 weeks training intervention. They will be randomized in one of the following three groups: poling specific motor skill training (10-12 x 3 repetitions maximum, RM) in specific designed cross country exercises 3 times per week in addition to their regular training. Further, maximal strength training in squat, dead lift, bench press, bench pull and pull down (2-5 x 3 repetitions RM) 3 times per week in addition to their regular training and a control group who only perform their regular training. Pre- and post intervention, all participants will perform tests in VO2max (running), VO2max (poling), work economy (poling), video and IMU analyzes of poling technique, time performance test (poling), motor skill tests and maximal strength tests.

ELIGIBILITY:
Inclusion Criteria:

* healthy, competitive cross country athletes 16-30 years old

Exclusion Criteria:

* contraindications to maximal strength training and strength and endurance testing

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Time trial poling on a roller ski tarmac track | 10 weeks
  Seconds used in a 6 km track.

SECONDARY OUTCOMES:
Video analyzes of technique | 10 weeks
  Joint angles. Unique outcome measure.
Analyzes of angular velocity by use of IMU (inertial movement devices) | 10 weeks
  Degree/second by use of gyrometer from the Musclelab System from Ergotest Technology. Unique outcome measure.
Analyzes of external force (N) in poles during poling | 10 weeks
  Force measurements by use of the Musclelab System from Ergotest Technology. Unique outcome measure.
Maximal pulldown strength (RM/kg) | 10 weeks
  Kilos in pulldown. Unique outcome measure.
Maximal leggpress strength (RM/kg) | 10 weeks
  Kilos in leggpress. Unique outcome measure.
Maximal pulldown power (Watt) | 10 weeks
  Watts in pulldown by use of Musclelab.System (Ergotest Technology). Unique outcome measure.
Maximal leggpress power (Watt) | 10 weeks
  Watts in leggpress by use of Musclelab.System (Ergotest Technology). Unique outcome measure.
Maximal oxygen uptake (VO2max, ml/kg/min) in running on treadmill | 10 weeks
  Ergospirometrical incremental (ramp) protocols using Cortex Metalyzer. Unique outcome measure.
Maximal oxygen uptake (VO2max, ml/kg/min) in poling on treadmill | 10 weeks
  Ergospirometrical incremental (ramp) protocols using Cortex Metalyzer. Unique outcome measure.
Lactate threshold (mmol/L blood) in poling on treadmill | 10 weeks
  Measurement of lactate using Lactate Scout (EKF Diagnostics) in different submaximal work periods up to the point reaching warm up values plus 2,3 mmol/L. Unique outcome measure.
Poling economy | 10 weeks
  Measurement of oxygen consumption per meter poling. Unique outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Arnstein Sunde, MSC, Principal Investigator — Telemark UC; Øyvind Støren, PhD, Study Chair — Telemark UC
Locations (1):
- Telemark UC, Bø, Telemark, Norway

IPD SHARING:
Plan to Share IPD: Yes
planned published in a peer reviewed journal

REFERENCES:
- [Background] Danielsen J, Sandbakk O, Holmberg HC, Ettema G. Mechanical Energy and Propulsion in Ergometer Double Poling by Cross-country Skiers. Med Sci Sports Exerc. 2015 Dec;47(12):2586-94. doi: 10.1249/MSS.0000000000000723. PMID 26110695
- [Background] Osteras H, Helgerud J, Hoff J. Maximal strength-training effects on force-velocity and force-power relationships explain increases in aerobic performance in humans. Eur J Appl Physiol. 2002 Dec;88(3):255-63. doi: 10.1007/s00421-002-0717-y. Epub 2002 Oct 17. PMID 12458369